CLINICAL TRIAL: NCT02875106
Title: BAYathlon - a Digital Non-interventional AF Screening Study to Identify Commercial Pulse Detection Systems (CPDS) Detecting AF and Sinus Rhythm Parallel to ECG Recording Within Routine Clinical Setting
Brief Title: A Digital Non-interventional Atrial Fibrillation (AF) Screening Study With Commercial Pulse Detection Systems
Acronym: BAYathlon
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18796
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Atrial Fibrillation
Keywords: Sinus rhythm
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Atrial Fibrillation Patients: Adult female and male patients with diagnosed atrial fibrillation
  Interventions: Device: 12-point-ECG; Device: Polar V800; Device: 360° eMotion FAROS SET + Belt; Device: Adidas Micoach smart run; Device: TomTom Runner Cardio HRM
- Sinus Rhythm Patients: Adult female and male patients with diagnosed sinus rhythm
  Interventions: Device: 12-point-ECG; Device: Polar V800; Device: 360° eMotion FAROS SET + Belt; Device: Adidas Micoach smart run; Device: TomTom Runner Cardio HRM

INTERVENTIONS:
Device: 12-point-ECG — routine recording will be 300 seconds
Device: Polar V800 — routine recording will be 300 seconds
Device: 360° eMotion FAROS SET + Belt — routine recording will be 300 seconds
Device: Adidas Micoach smart run — routine recording will be 300 seconds
Device: TomTom Runner Cardio HRM — routine recording will be 300 seconds

SUMMARY:
The primary objective in this study is to identify commercial pulse detection systems (CPDS) parallel to electrocardiogram (ECG) recording within routine clinical setting, which are able to detect atrial fibrillation or sinus rhythm of screened patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult female and male patients for whom the decision to record an ECG was made as per investigator's routine treatment practice
* Patient able and willing to provide signed informed consent

Exclusion Criteria:

* Patients with any comorbidities or abnormalities of heart function or rhythm, which might, in the opinion of the investigator, interfere with the evaluation of study data
* Patients participating in an investigational program with interventions outside of routine clinical practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients for whom the decision to record an ECG was made as per investigator's routine treatment practice
Sampling Method: Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-05-08 (Actual)

PRIMARY OUTCOMES:
The rate of correctly detected atrial fibrillation signals by CPDS in reference to ECG (sensitivity of CPDS). | 120 seconds
  This will be calculated as proportion of patients with atrial fibrillation diagnosed by CPDS record out of the total number of patients diagnosed with atrial fibrillation by ECG record (for patients with diagnosis for both recordings available).

SECONDARY OUTCOMES:
The rate of correctly detected sinus rhythm signals by CPDS in reference to ECG (sensitivity of CPDS). | 120 seconds
  This will be calculated as proportion of patients with sinus rhythm diagnosed by CPDS record out of the total number of patients diagnosed with sinus rhythm by ECG record (for patients with diagnosis for both recordings available).
The rate of correctly detected AF of the applied algorithm of the ECG-data in reference to the primary diagnosis of the investigator using the ECG-graph (sensitivity of algorithm). | 120 seconds
  This will be calculated as proportion of AF patients detected by the applied algorithm compared with proportion of AF patients diagnosed by the investigator, both based on ECG records.
The rate of correctly detected atrial fibrillation signals by CPDS in reference to ECG (sensitivity of CPDS). | 60 seconds, 180 seconds, 240 seconds, 300 seconds
  This will be a sensitivity analysis of derived sensitivities of CPDS in different time frames, calculated as proportion of patients with sinus rhythm diagnosed by CPDS record out of the total number of patients diagnosed with sinus rhythm by ECG record (for patients with diagnosis for both recordings available).

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Multiple Locations, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] Muller C, Hengstmann U, Fuchs M, Kirchner M, Kleinjung F, Mathis H, Martin S, Blase I, Perings S. Distinguishing atrial fibrillation from sinus rhythm using commercial pulse detection systems: The non-interventional BAYathlon study. Digit Health. 2021 May 22;7:20552076211019620. doi: 10.1177/20552076211019620. eCollection 2021 Jan-Dec. PMID 34104466
- See also: Related Info — http://clinicaltrials.bayer.com